CLINICAL TRIAL: NCT07027696
Title: Sexual Health of Women With Genital Mutilation Seen at the Saint-Denis Women's Center
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0061_MAISON DES FEMMES
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Female Genital Mutilation; Sexual Dysfunctions, Psychological; Sexual Health; Violence Against Women; Post-Traumatic Stress Disorders; Acculturation; Women's Health Services; Refugees
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at the sexual health of women who have experienced female genital mutilation (FGM) and who are receiving care at the Women's Center at Saint-Denis Hospital. It aims to better understand their sexual experiences, including the impact of past violence and trauma, and to explore how multidisciplinary care (such as psychological and sexological support) can help. The study also looks at what women expect from their care and how they feel about surgical or other types of support.

ELIGIBILITY:
Inclusion Criteria:

* Women with female genital mutilation (FGM), or considered to be excised, consulting at the Maison des Femmes (Women's House) at Saint-Denis Hospital.
* Women enrolled in the multidisciplinary care pathway for FGM.

Exclusion Criteria:

- Women under the age of 15.

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult women who have experienced female genital mutilation (FGM) or are considered to be excised, and who are consulting at the Maison des Femmes (Women's House) of the Saint-Denis Hospital in France. These women are engaged in a multidisciplinary care pathway addressing the consequences of FGM. Most are migrants who have faced various forms of violence, either in their country of origin or during their migration journey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the sexual function profile of women with female genital mutilation (FGM) during consensual sexual activity, using a structured clinical sexological evaluation that accounts for histories of violence. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France